CLINICAL TRIAL: NCT03030638
Title: Drug Utilization Study for Olodaterol
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: RTI health solutions, US (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1222.53
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; indacaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Olodaterol: Patients initiating Olodaterol for the first time
  Interventions: Drug: Olodaterol
- Indacaterol: Patients initiating Indacaterol for the first time
  Interventions: Drug: Indacaterol

INTERVENTIONS:
Drug: Olodaterol — Drug
  Other Names: STRIVERDI
  Groups: Olodaterol
Drug: Indacaterol — Drug
  Groups: Indacaterol

SUMMARY:
This study aims to characterise the use of single-agent olodaterol and single-agent indacaterol, the only marketed long-acting beta2-agonist (LABA)s authorised for chronic obstructive pulmonary disease (COPD), but not for asthma, in clinical practice.

DETAILED DESCRIPTION:
Boehringer Ingelheim GmbH (BI) developed olodaterol, an inhaled long-acting beta2-agonist (LABA), for the indication of chronic obstructive pulmonary disease (COPD). Because the use of LABAs has been associated with increased morbidity and mortality in patients with asthma, the health authorities requested the conduct of a post-approval drug utilisation study to assess potential off-label use of olodaterol in asthma and to characterise the use of olodaterol in clinical practice. The single agent indacaterol, the only other marketed LABA authorised in clinical practice for COPD but not for asthma, will also be assessed. Study objectives include the following: (1) Quantify the frequency of off-label use of olodaterol and indacaterol among new users of these medications; and (2) Describe the baseline characteristics of new users of olodaterol and indacaterol. This cross-sectional study will use information among new users of olodaterol or indacaterol collected in the following healthcare databases: the PHARMO Database Network in the Netherlands, the National Registers in Denmark, and the IMS Health Information Solutions (IMS) Real-World Evidence (RWE) Longitudinal Patient Database (LPD) in France. The source population is all patients enrolled in the selected study databases at the date olodaterol became available in each database's country. The study groups are those patients from the source population who receive a first dispensing for single-agent formulations of olodaterol for the primary objective or indacaterol for the secondary objective and have at least 12 months of continuous enrolment in the study databases. The study will describe the number and proportion of new users by indication and potential off-label use and according to medical history and use of co-medications.

ELIGIBILITY:
Inclusion criteria:

* receive a first prescription/dispensing for single-agent formulations of olodaterol or indacaterol during the study period (no prescriptions/dispensings ever before)
* patients must have at least 12 consecutive months of enrolment in the database before the index date

Exclusion criteria:

- Individuals with missing or implausible values for age or sex will be excluded.

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study source population includes all patients enrolled in the selected study databases at the date both olodaterol and indacaterol are available in each database's country. The study is planned to be conducted in the following databases: the PHARMO Database Network in the Netherlands, the National Registers in Denmark, and the Real-World Evidence (RWE) Longitudinal Patient Database (LPD) in France.
Sampling Method: Probability Sample
Enrollment: 27606 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Aarhus Universitetshospital Skejby, Aarhus, Denmark
- IMS Health Information solutions, Courbevoie, France
- Pharmo Institute, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited in the study are those patients who received a first dispensing for single-agent formulations of olodaterol or indacaterol during the study period and had at least 12 months of continuous enrolment in the study databases prior to index date.
Pre-assignment Details: Databases used: PHARMO Database Network in the Netherlands, National Registers in Denmark and IMS Health Information Solutions Real-World Evidence (RWE) Longitudinal Patient Database (LPD) in France. Study periods were 01 March 2014 - 31 December 2016 in PHARMO and Denmark and 01 October 2015 - 30 November 2017 in the IMS RWE LPD panels.
Groups:
- Olodaterol - PHARMO Overall: Patients from the data source PHARMO overall received Olodaterol inhalation solution via Striverdi Respimat inhaler for the first time, continuing for 12 months.
- Indacaterol - PHARMO Overall: Patients from the data source PHARMO overall received Indacaterol inhalation powder for the first time, continuing for 12 months.
- Olodaterol - National Health Databases, Denmark: Patients from the data source National Health Databases, Denmark received Olodaterol inhalation solution via Striverdi Respimat inhaler for the first time, continuing for 12 months.
- Indacaterol - National Health Databases, Denmark: Patients from the data source National Health Databases, Denmark received Indacaterol inhalation powder for the first time, continuing for 12 months.
- Olodaterol - IMS RWE LPD General Practitioner (GP) Panel: Patients from the data source IMS RWE LPD GP panel received Olodaterol inhalation solution via Striverdi Respimat inhaler for the first time, continuing for 12 months.
- Indacaterol - IMS RWE LPD GP Panel: Patients from the data source IMS RWE LPD GP Panel received Indacaterol inhalation powder for the first time, continuing for 12 months.
- Olodaterol - IMS RWE LPD Pulmonologist Panel: Patients from the data source IMS RWE LPD pulmonologist panel received Olodaterol inhalation solution via Striverdi Respimat inhaler for the first time, continuing for 12 months.
- Indacaterol - IMS RWE LPD Pulmonologist Panel: Patients from the data source IMS RWE LPD Pulmonologist Panel received Indacaterol inhalation powder for the first time, continuing for 12 months.
Period: Overall Study
Arm/Group | Olodaterol - PHARMO Overall | Indacaterol - PHARMO Overall | Olodaterol - National Health Databases, Denmark | Indacaterol - National Health Databases, Denmark | Olodaterol - IMS RWE LPD General Practitioner (GP) Panel | Indacaterol - IMS RWE LPD GP Panel | Olodaterol - IMS RWE LPD Pulmonologist Panel | Indacaterol - IMS RWE LPD Pulmonologist Panel
Started | 1386 | 1841 | 1712 | 6406 | 696 | 1592 | 364 | 127
PHARMO-GP (Sub-set of PHARMO Overall) | 372 | 636 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1386 | 1841 | 1712 | 6406 | 696 | 1592 | 364 | 127
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population: The study population included those patients from the source population who received a first dispensing for single-agent formulations of olodaterol or indacaterol during the study period and had at
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol - PHARMO Overall | Indacaterol - PHARMO Overall | Olodaterol - National Health Databases, Denmark | Indacaterol - National Health Databases, Denmark | Olodaterol - IMS RWE LPD General Practitioner (GP) Panel | Indacaterol - IMS RWE LPD GP Panel | Olodaterol - IMS RWE LPD Pulmonologist Panel | Indacaterol - IMS RWE LPD Pulmonologist Panel | Total
Number analyzed (Participants) | 1386 | 1841 | 1712 | 6406 | 696 | 1592 | 364 | 127 | 14124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.9 (11.33) | 66.3 (12.83) | 70.6 (11.12) | 68.3 (11.45) | 62.5 (13.77) | 62.4 (14.40) | 65.8 (13.26) | 67.3 (13.39) | 67.2 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 702 | 887 | 977 | 3324 | 322 | 696 | 129 | 42 | 7079
  Male | 684 | 954 | 735 | 3082 | 374 | 896 | 235 | 85 | 7045
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Off-label Use of Olodaterol Among New Users
Description: Percentage of off-label use of olodaterol among new users of this medication. Potential off-label are the patients, aged 18 years or older with no recorded Chronic Obstructive Pulmonary Disease (COPD) diagnosis and no asthma diagnosis. Off-label are the patients, aged 17 years or younger or patients aged 18 years or older with no recorded COPD diagnosis but with a diagnosis of asthma. Index date is defined as the date an eligible patient receives the first dispensing of olodaterol or indacaterol during the study period.
Time Frame: 01March2014 to 30November2017 up to 30 days after index date, up to 1370 days.
Population: Study population
Measure: Number; unit: Percentage of participants
Groups:
- Olodaterol - PHARMO-GP: Patients from the data source PHARMO-GP received Olodaterol inhalation solution via Striverdi Respimat inhaler for the first time, continuing for 12 months.
Arm/Group | Olodaterol - PHARMO Overall | Olodaterol - PHARMO-GP | Olodaterol - National Health Databases, Denmark | Olodaterol - IMS RWE LPD General Practitioner (GP) Panel | Olodaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1386 | 372 | 1712 | 696 | 364
Percentage of participants
  Potential off-label | 48.6 | 19.6 | 30.3 | 33.9 | 17.3
  Off-label | 3.5 | 6.2 | 4.4 | 12.4 | 4.9

2. Secondary Outcome: Percentage of Off-label Use of Indacaterol Among New Users
Description: Percentage of off-label use of Indacaterol among new users of this medication. Potential off-label are the patients, aged 18 years or older with no recorded COPD diagnosis and no asthma diagnosis. Off-label are the patients, aged 17 years or younger or patients aged 18 years or older with no recorded COPD diagnosis but with a diagnosis of asthma.
Time Frame: 01March2014 to 30November2017 up to 30 days after index date, up to 1370 days.
Population: Study population
Measure: Number; unit: Percentage of participants
Groups:
- Indacaterol - PHARMO-GP: Patients from the data source PHARMO-GP received Indacaterol inhalation powder for the first time, continuing for 12 months.
Arm/Group | Indacaterol - PHARMO Overall | Indacaterol - PHARMO-GP | Indacaterol - National Health Databases, Denmark | Indacaterol - IMS RWE LPD GP Panel | Indacaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1841 | 636 | 6406 | 1592 | 127
Percentage of participants
  Potential off-label | 61.1 | 29.2 | 66.6 | 34.9 | 20.5
  Off-label | 3.5 | 6.8 | 4.6 | 11.9 | 9.4

3. Secondary Outcome: Baseline Characteristics of New Users of Indacaterol: Age
Description: Baseline characteristics of patients in treatment group by data source: Age
Time Frame: Baseline
Population: Study population
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Indacaterol - PHARMO Overall | Indacaterol - National Health Databases, Denmark | Indacaterol - IMS RWE LPD GP Panel | Indacaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1841 | 6406 | 1592 | 127
Years | 67 [59.0 to 75.0] | 69 [61.2 to 76.5] | 63 [53.0 to 73.0] | 68 [59.0 to 78.0]

4. Primary Outcome: Baseline Characteristics of New Users of Olodaterol: Age
Description: Baseline characteristics of patients in treatment group by data source: Age
Time Frame: Baseline
Population: Study population
Measure: Median (Inter-Quartile Range); unit: Years
Arm/Group | Olodaterol - PHARMO Overall | Olodaterol - National Health Databases, Denmark | Olodaterol - IMS RWE LPD General Practitioner (GP) Panel | Olodaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1386 | 1712 | 696 | 364
Years | 68 [60.0 to 75.0] | 71 [64.0 to 78.5] | 63 [53.0 to 72.0] | 67 [59.0 to 75.0]

5. Primary Outcome: Baseline Characteristics of New Users of Olodaterol: Gender
Description: Baseline characteristics of patients in treatment group by data source: Gender
Time Frame: Baseline
Population: Study population
Measure: Count of Participants; unit: Participants
Arm/Group | Olodaterol - PHARMO Overall | Olodaterol - National Health Databases, Denmark | Olodaterol - IMS RWE LPD General Practitioner (GP) Panel | Olodaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1386 | 1712 | 696 | 364
Participants
  Female | 702 | 977 | 322 | 129
  Male | 684 | 735 | 374 | 235

6. Secondary Outcome: Baseline Characteristics of New Users of Indacaterol: Gender
Description: Baseline characteristics of patients in treatment group by data source: Gender
Time Frame: Baseline
Population: Study population
Measure: Count of Participants; unit: Participants
Arm/Group | Indacaterol - PHARMO Overall | Indacaterol - National Health Databases, Denmark | Indacaterol - IMS RWE LPD GP Panel | Indacaterol - IMS RWE LPD Pulmonologist Panel
Number analyzed (Participants) | 1841 | 6406 | 1592 | 127
Participants
  Female | 887 | 3324 | 696 | 42
  Male | 954 | 3082 | 896 | 85

ADVERSE EVENTS:
Time Frame: Based on the data planned for this study, no suspected adverse events/reactions were expected.
Description: Adverse Events were not monitored/assessed
Arm/Group | Olodaterol | Indacaterol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-02-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03030638/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03030638/SAP_001.pdf